CLINICAL TRIAL: NCT05772832
Title: COMPARISON OF DEXMEDETOMIDINE AND REMIFENTANIL FOR POSTOPERATIVE PAIN IN TRANSPHENOIDAL Pituitary SURGERY
Status: Completed | Type: Observational
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, İpek İZGİN AVCI, principal investigator, Kocaeli University
Other Study IDs: KocaeliUI
Record Dates: First submitted 2023-02-18; First posted 2023-03-16 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Postoperative Pain
Keywords: DEXMEDETOMİDİNE; REMİFENTANYL; pituitary SURGERY
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexmedetomidine; Remifentanil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- GROUP USING REMIFENTANYL: THE GROUP USING PEROPERATIVE REMIFENTANYL AND PROPOFOL IN TRANSSPHENOIDAL Pituitary Surgery 0.01-0.2 μg /kg /min Remifentanyl and 3-12 mg/kg/h propofol
  Interventions: Drug: Remifentanyl
- GROUP USING DEXMEDETOMIDINE: THE GROUP USING PEROPERATIVE DEXMEDETOMIDINE AND PROPOFOL IN TRANSSPHENOIDAL Pituitary Surgery 0.01-0.02 μg/kg/min (~0.5 μg/kg/h) continuous infusion of dexmedetomidine 1 mcg/kg 10 minutes after a loading dose and 3-12 mg/kg/h propofol
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Efficacy of dexmedetomidine on postoperative pain in patients undergoing transsphenoidal pituitary surgery
  Groups: GROUP USING DEXMEDETOMIDINE
Drug: Remifentanyl — Efficacy of remifentanyl on postoperative pain in patients undergoing transsphenoidal pituitary surgery
  Groups: GROUP USING REMIFENTANYL

SUMMARY:
In patients with pituitary adenoma scheduled for endoscopic transsphenoidal pituitary surgery, it was aimed to compare the efficacy of postoperative pain relief of a selective α-2 agonist "Dexmedetomidine" and the rapid and short-acting opioid "Remifentanil" using the "Numerical Rating Scale" (NRS) administered alongside propofol in perioperative maintenance anesthesia. .

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* ASA-1 and ASA-2 patients

Exclusion Criteria:

* Patients in need of postoperative intensive care

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing transsphenoidal pituitary surgery
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2023-02-22 (Actual)

PRIMARY OUTCOMES:
postoperative pain scale | at post anesthesia care unit (T1)
  Comparison of postoperative Numerical Rating Scale(NRS) values of both study arms(min 0, max 10; 10 is unbearable pain )
postoperative pain scale | 2 hours after surgery (T2)
  Comparison of postoperative Numerical Rating Scale(NRS) values of both study arms(min 0, max 10; 10 is unbearable pain )
postoperative pain scale | 8 hours after surgery (T3)
  Comparison of postoperative Numerical Rating Scale(NRS) values of both study arms(min 0, max 10; 10 is unbearable pain )
postoperative pain scale | 24 hours after surgery (T4)
  Comparison of postoperative Numerical Rating Scale(NRS) values of both study arms(min 0, max 10; 10 is unbearable pain )

SECONDARY OUTCOMES:
need for analgesics | Additional analgesic drug requirements at post anesthesia care unit (T1)
  Comparison of whether there is a need for additional POSTOPERATIVE analgesic medication
need for analgesics | Additional analgesic drug requirements at 2 hours after surgery (T2)
  Comparison of whether there is a need for additional POSTOPERATIVE analgesic medication
need for analgesics | Additional analgesic drug requirements at 8 hours after surgery (T3)
  Comparison of whether there is a need for additional POSTOPERATIVE analgesic medication
need for analgesics | Additional analgesic drug requirements at 24 hours after surgery (T4)
  Comparison of whether there is a need for additional POSTOPERATIVE analgesic medication
Comparison of postoperative nausea-vomiting rate | at post anesthesia care unit (T1)
  Comparison of postoperative nausea-vomiting rate
Comparison of postoperative nausea-vomiting rate | 2 hours after surgery (T2)
  Comparison of postoperative nausea-vomiting rate
Comparison of postoperative nausea-vomiting rate | 8 hours after surgery (T3)
  Comparison of postoperative nausea-vomiting rate
Comparison of postoperative nausea-vomiting rate | 24 hours after surgery (T4)
  Comparison of postoperative nausea-vomiting rate

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kocaeli, Kocaeli, IZMIT, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zheng Y, Cui S, Liu Y, Zhang J, Zhang W, Zhang J, Gu X, Ma Z. Dexmedetomidine prevents remifentanil-induced postoperative hyperalgesia and decreases spinal tyrosine phosphorylation of N-methyl-d-aspartate receptor 2B subunit. Brain Res Bull. 2012 Mar 10;87(4-5):427-31. doi: 10.1016/j.brainresbull.2012.01.009. Epub 2012 Jan 25. PMID 22301064
- [Background] Lee C, Kim YD, Kim JN. Antihyperalgesic effects of dexmedetomidine on high-dose remifentanil-induced hyperalgesia. Korean J Anesthesiol. 2013 Apr;64(4):301-7. doi: 10.4097/kjae.2013.64.4.301. Epub 2013 Apr 22. PMID 23646238
- [Background] Venn RM, Hell J, Grounds RM. Respiratory effects of dexmedetomidine in the surgical patient requiring intensive care. Crit Care. 2000;4(5):302-8. doi: 10.1186/cc712. Epub 2000 Jul 31. PMID 11056756
- [Background] Virtanen R, Savola JM, Saano V, Nyman L. Characterization of the selectivity, specificity and potency of medetomidine as an alpha 2-adrenoceptor agonist. Eur J Pharmacol. 1988 May 20;150(1-2):9-14. doi: 10.1016/0014-2999(88)90744-3. PMID 2900154
- [Background] Hwang W, Lee J, Park J, Joo J. Dexmedetomidine versus remifentanil in postoperative pain control after spinal surgery: a randomized controlled study. BMC Anesthesiol. 2015 Feb 24;15:21. doi: 10.1186/s12871-015-0004-1. eCollection 2015. PMID 25750586
- [Background] Javaherforooshzadeh F, Monajemzadeh SA, Soltanzadeh M, Janatmakan F, Salari A, Saeed H. A Comparative Study of the Amount of Bleeding and Hemodynamic Changes between Dexmedetomidine Infusion and Remifentanil Infusion for Controlled Hypotensive Anesthesia in Lumbar Discopathy Surgery: A Double-Blind, Randomized, Clinical Trial. Anesth Pain Med. 2018 Apr 28;8(2):e66959. doi: 10.5812/aapm.66959. eCollection 2018 Apr. PMID 30009153
- [Background] Rajan S, Hutcherson MT, Sessler DI, Kurz A, Yang D, Ghobrial M, Liu J, Avitsian R. The Effects of Dexmedetomidine and Remifentanil on Hemodynamic Stability and Analgesic Requirement After Craniotomy: A Randomized Controlled Trial. J Neurosurg Anesthesiol. 2016 Oct;28(4):282-90. doi: 10.1097/ANA.0000000000000221. PMID 26325514
- [Background] Choi EK, Seo Y, Lim DG, Park S. Postoperative nausea and vomiting after thyroidectomy: a comparison between dexmedetomidine and remifentanil as part of balanced anesthesia. Korean J Anesthesiol. 2017 Jun;70(3):299-304. doi: 10.4097/kjae.2017.70.3.299. Epub 2017 Mar 15. PMID 28580080
- [Background] Ge DJ, Qi B, Tang G, Li JY. Intraoperative Dexmedetomidine Promotes Postoperative Analgesia and Recovery in Patients after Abdominal Colectomy: A CONSORT-Prospective, Randomized, Controlled Clinical Trial. Medicine (Baltimore). 2015 Oct;94(43):e1727. doi: 10.1097/MD.0000000000001727. PMID 26512563
- [Background] Salman N, Uzun S, Coskun F, Salman MA, Salman AE, Aypar U. Dexmedetomidine as a substitute for remifentanil in ambulatory gynecologic laparoscopic surgery. Saudi Med J. 2009 Jan;30(1):77-81. PMID 19139778
- [Background] Hamed JME, Refaat HSM, Al-Wadaani H. Dexmedetomidine Compared to Remifentanil Infusion as Adjuvant to Sevoflurane Anesthesia during Laparoscopic Sleeve Gastrectomy. Anesth Essays Res. 2019 Oct-Dec;13(4):636-642. doi: 10.4103/aer.AER_126_19. Epub 2019 Dec 16. PMID 32009708